CLINICAL TRIAL: NCT04056611
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Clinical Outcomes, Antiviral Activity, Safety, Tolerability, Pharmacokinetics, and Pharmacokinetics/Pharmacodynamics of JNJ-53718678 in Adult and Adolescent Hematopoietic Stem Cell Transplant Recipients With Respiratory Syncytial Virus Infection of the Upper Respiratory Tract
Brief Title: Effects of JNJ-53718678 in Adult and Adolescent Participants Who Had a Hematopoietic Stem Cell Transplantation and Who Are Infected With Respiratory Syncytial Virus (RSV)
Acronym: FREESIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A strategic decision was made to discontinue the study. The decision was not based on a safety concern.
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108662; 53718678RSV2005 (Other: Janssen Sciences Ireland UC); 2019-001551-39 (EudraCT Number)
Expanded Access: NCT04221412 (No longer available)
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult cohort: JNJ-53718678 or Placebo (Experimental): Participants greater than or equal to (>=) 18 to less than or equal to (<=) 75 years of age will receive 250 milligram (mg) JNJ-53718678 twice daily (bid) for 21 days (without coadministration with moderate or strong CYP3A4 inhibitors), or 125 mg JNJ-53718678 bid for 21 days (coadministered with moderate or strong CYP3A4 inhibitors with the exception of posaconazole), or 125 mg once daily (qd) for 21 days (when coadministered with posaconazole), or matching placebo for 21 days.
  Interventions: Drug: JNJ-53718678 250 mg; Drug: Placebo; Drug: JNJ-53718678 125 mg
- Adolescent cohort: JNJ-53718678 or Placebo (Experimental): Participants >=13 to <18 years of age will receive 250 mg JNJ-53718678 bid for 21 days (without coadministration with moderate or strong CYP3A4 inhibitors), or 125 mg JNJ-53718678 bid for 21 days (coadministered with moderate or strong CYP3A4 inhibitors with the exception of posaconazole), or 125 mg qd for 21 days (when coadministered with posaconazole), or matching placebo for 21 days.
  Interventions: Drug: JNJ-53718678 250 mg; Drug: Placebo; Drug: JNJ-53718678 125 mg

INTERVENTIONS:
Drug: JNJ-53718678 250 mg — JNJ-53718678 250 mg will be administered orally.
Drug: Placebo — Matching placebo will be administered orally.
Drug: JNJ-53718678 125 mg — JNJ-53718678 125 mg will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the effect of JNJ-53718678 on the development of respiratory syncytial virus (RSV) lower respiratory tract infection (LRTIs) in adult hematopoietic stem cell transplant (HSCT) recipients with RSV upper RTI.

DETAILED DESCRIPTION:
RSV is recognized as major respiratory pathogen in infants and young children and causes upper and lower respiratory illness among all age groups, often going undiagnosed. Immunocompromised (IC) participants have a reduced ability to combat infection due to an impaired or weakened immune system. Within the IC population, HSCT recipients are generally regarded as having a particularly high risk for more severe disease caused by RSV, representing a substantial unmet need for antiviral treatment of RSV infections in this participant population. JNJ-53718678 is an investigational, potent, small molecule, respiratory syncytial virus (RSV)-specific fusion inhibitor. The study will include a Screening Period (Day -2 to Day 1), a Treatment Period (Day 1 to Day 21), and a Follow-up Period (1 year). Assessments like chest X-ray, pulse/heart rate, respiratory rate, electrocardiogram (ECG), etc will be performed. Safety and efficacy will be assessed through the study. The total study duration for each participant will be approximately 49 days.

ELIGIBILITY:
Inclusion Criteria:

* Received an autologous or allogeneic hematopoietic stem cell transplant (HSCT) using any conditioning regimen
* Absolute lymphocyte count (ALC) less than (<) 1,000 cells/microliter (mL)
* Participant has laboratory confirmed RSV diagnosis within 48 hours of randomization
* New onset of at least 1 of the following respiratory symptoms within 4 days prior to the anticipated start of dosing nasal congestion, rhinorrhea, cough or pharyngitis (sore throat), and/or worsening of one of these chronic (associated with previously existing diagnosis, example, chronic rhinorrhea, seasonal allergies, chronic lung disease) respiratory symptoms within 4 days prior to the anticipated start of dosing
* Peripheral capillary oxygen saturation (SpO2) greater than or equal to (>=) 92 percent (%) on room air

Exclusion Criteria:

* Admitted to the hospital primarily for a lower respiratory tract disease of any cause as determined by the investigator
* Requires supplemental oxygen at Screening or any time between Screening and randomization
* Documented to be positive for other respiratory viruses (limited to influenza, parainfluenza, human rhinovirus, adenovirus, human metapneumovirus, or coronavirus) within 7 days prior to or at the Screening visit, if determined by local SOC testing (additional testing is not required)
* Clinically significant bacteremia or fungemia within 7 days prior to or at Screening that has not been adequately treated, as determined by the investigator

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (69):
- United States (9):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Henry Ford Hospital - Hematology/oncology, Detroit, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Northwell Health Cancer Institute, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Baylor Scott and White Research Institute, Dallas, Texas
  - MD Anderson Cancer Center - University of Texas, Houston, Texas
- Argentina (5):
  - Hospital Espanol De Bahia Blanca, Bahía Blanca
  - Hospital Italiano de La Plata, Ciudad de La Plata
  - Sanatorio Allende, Córdoba
  - Hospital Privado-Universitario de Cordoba, Córdoba
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - Westmead Hospital, Westmead
- Belgium (7):
  - AZ Sint-Jan, Bruges
  - Jules Bordet Institute, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU de Liege, Liège
  - Jessa Ziekenhuis, Limbourg
- Brazil (10):
  - Fundacao Pio XII, Barretos
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Universidade Federal do Ceara Hospital Universitario Walter Cantidio, Fortaleza
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Sociedade Beneficente de Senhoras - Hospital Sírio Libanês, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- Bulgaria (3):
  - UMHAT 'Sveti Georgi'-Plovdiv, Plovdiv
  - Specialized Hospital for Active Treatment of Haematologic Diseases, Sofia
  - Multiprofile Hospital for Active Treatment 'Sveta Marina' EAD, Varna
- France (2):
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky (Ichilov) Medical Center, Tel Aviv
- Italy (2):
  - Ospedale San Raffaele HSR Istituto Scientifico Universitario San Raffaele, Milan
  - Ematologia Fondazione Univ. Policlinico Gemelli Università Cattolica del Sacro Cuore, Roma
- Japan (5):
  - Akita University Hospital, Akita
  - Chiba University Hospital, Chiba
  - Tokai University Hospital, Isehara
  - Japanese Red Cross Society Nagano Hospital, Nagano
  - Okayama University Hospital, Okayama
- Malaysia (4):
  - Hospital Ampang, Ampang
  - Penang General Hospital, George Town
  - University Malaya Medical Centre, Kuala Lumpur
  - Sunway Medical Centre, Petaling Jaya
- Leiden University Medical Center, Leiden, Netherlands
- The Catholic University of Korea Seoul St Mary s Hospital, Seoul, South Korea
- Spain (7):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
- Skanes universitetssjukhus, Malmo, Sweden
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Kings College Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive either rilematovir or placebo. The dose was dependent upon coadministration without/with CYP3A4 inhibitors or posaconazole. Due to the limited participants randomized and due to chance, no participants were randomized to placebo.
Groups:
- JNJ-53718678: Participants with age greater than or equal to (>=) 18 to less than or equal to (<=) 75 years received rilematovir 125 milligrams (mg) twice daily (bid) for 21 days.
Period: Overall Study
Arm/Group | JNJ-53718678
Started | 3
Completed | 2
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 1
  FRANCE | 1
  ISRAEL | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Infection (LRTI)
Description: Percentage of participants who developed RSV LRTI was assessed. RSV LRTI was defined as the development of a lower respiratory sign or symptom (including decrease in oxygen saturation or increase in supplemental oxygen to maintain oxygen saturation, wheezing, rhonchi, rales, dyspnea, tachypnea, worsening cough) and positive RSV test from lower respiratory tract sample (example [eg], sputum, induced sputum, bronchoalveolar lavage (BAL), lung biopsy, or autopsy specimen) within +-4 days of a new chest image finding, compared to baseline, consistent with a LRTI; OR positive RSV test from lower respiratory tract sample (eg, sputum, induced sputum, BAL, lung biopsy, or autopsy specimen) only; OR positive RSV test from upper respiratory tract sample within ±4 days of a new chest image finding, compared to baseline, consistent with a RSV LRTI as determined by the Endpoint Adjudication Committee (EAC).
Time Frame: Up to Day 28
Population: Efficacy analysis set included all participants who were randomized, treated (took at least 1 dose), and had a RSV infection confirmed by central laboratory analysis, excluding participants infected with a co-pathogen at baseline not identified during screening, analyzed as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

2. Secondary Outcome: Percentage of Participants Who Developed RSV-associated Lower Respiratory Tract Complication (LRTC)
Description: Percentage of participants who developed RSV-associated LRTC was assessed. RSV-associated LRTC defined as development of lower respiratory sign/symptom (includes decrease in oxygen saturation/increase in supplemental oxygen to maintain oxygen saturation, wheezing, rhonchi, rales, dyspnea, tachypnea, and worsening cough) and met 1 of following subcategories determined by EAC: a) RSV LRTI, b) secondary bacterial LRTI (positive specimen for clinically significant bacterium within 4 days of new chest image finding, compared to baseline, consistent with LRTI), c) secondary LRTI due to unusual pathogens (positive specimen for clinically significant unusual organism within 4 days of new chest image finding, compared to baseline, consistent with LRTI), d) secondary LRTC of unknown etiology (new chest image finding than baseline, consistent with LRTI, inflammatory process/ some other clinically significant pulmonary process which were absent within 4 days of new chest image finding).
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the intervention. Any AE which occurred post first dose administration of study drug up to the end of study (EOS) (that is, Day 49) was considered as treatment-emergent.
Time Frame: Up to Day 49
Population: The safety analysis set included all randomized participants who took at least 1 dose of study intervention and were analyzed 'as treated'.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Participants | 2

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Abnormal (>=Grade 3) Clinical Laboratory Findings
Description: Percentage of participants with greater than or equal to (>=) Grade 3 treatment-emergent laboratory abnormalities (platelet count decreased, glucose increase) was assessed in this outcome measure. Treatment-emergent: any abnormality occurred post first dose of study drug up to end of study (that is, Day 49).
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants
  Platelet count decreased | 33.33
  Glucose increase | 33.33

5. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Findings
Description: Percentage of participants with clinically significant abnormalities in ECG findings was assessed in this outcome measure. Various ECG variables assessed were heart rate: abnormally low (<= 45 beats per minute [bpm]), abnormally high (>= 120 bpm); PR interval: abnormally high (>=210 milliseconds [msec]); QRS interval: abnormally high (>=120 msec), QT interval and corrected QT (QTcF; according to Fridericia's formula) interval (>450 msec, >480 msec, or >500 msec, increases from baseline >30 msec or >60 msec.)
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants
  Heart rate | 0
  PR interval | 0
  QRS interval | 0
  QTcF | 0

6. Secondary Outcome: Percentage of Participants With Treatment-emergent Abnormal Vital Signs Findings
Description: Percentage of participants with abnormal vital signs findings was assessed. Abnormal vital parameters included pulse rate: abnormally low <=45 bpm, abnormally high >=120 bpm; Systolic Blood Pressure (SBP): abnormally low <=90 Millimeter of mercury (mmHg), Grade 1 (mild): > 90 mmHg - < 100 mmHg, Grade 2 (moderate): >= 100 mmHg to <110 mmHg, Grade 3 (severe): >=110 mmHg; Diastolic BP: abnormally low <=50 mmHg, Grade 1: >90 mmHg to <100 mmHg, Grade 2: >=100 mmHg to <110 mmHg, Grade 3: >=110 mmHg; Respiratory rate- Grade 1 (mild): 17-20 breaths per minute, Grade 2 (moderate): 21-25 breaths per minute, Grade 3 (severe): >25 breaths per minute, Grade 4 (potentially life threatening): intubation; Temperature: abnormally high >38.0 degree celsius. Vital signs abnormalities reported for at least 1 participant were reported in this outcome measure. Treatment-emergent: any abnormality occurred post first dose of study drug up to EOS (that is, Day 49).
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants
  Respiratory rate: Grade 2 | 66.67
  DBP: Grade 1 | 33.3

7. Secondary Outcome: Percentage of Participants Who Progressed to Respiratory Failure (of Any Cause) Requiring Mechanical Ventilation (Invasive or Noninvasive) and/or Death Among Those Who Developed RSV LRTI or RSV-associated LRTC Per the EAC's Assessment
Description: Percentage of participants who progressed to respiratory failure (of any cause) requiring mechanical ventilation (invasive or noninvasive) and/or death among those who developed RSV LRTI or RSV-associated LRTC per the EAC's assessment was assessed. Here, '0' in the 'number of participants analyzed' field (N=0) signifies that no participants were available for the analysis because none of the participants developed RSV LRTI or RSV-associated LRTC per the EAC's Assessment.
Time Frame: Up to Day 49
Population: as for outcome 1
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage of Participants Who Progressed to Respiratory Failure (of Any Cause) Requiring Mechanical Ventilation (Invasive or Noninvasive) and/or Death (All-cause Mortality)
Description: Percentage of participants who progressed to respiratory failure (of any cause) requiring mechanical ventilation (invasive or noninvasive) and/or death (all-cause mortality) was assessed.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

9. Secondary Outcome: Percentage of Participants Who Progressed to Death (All-cause Mortality) Among Those Who Developed RSV LRTI or RSV-associated LRTC Per the EAC's Assessment
Description: Percentage of participants who progressed to death (all-cause mortality) among those who developed RSV LRTI or RSV-associated LRTC per the EAC's assessment was assessed. Here, '0' in the 'number of participants analyzed' field (N=0) signifies that no participants were available for the analysis because none of the participants developed RSV LRTI or RSV-associated LRTC per the EAC's Assessment.
Time Frame: Up to Day 49
Population: as for outcome 1
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants Who Progressed to Death (All-cause Mortality)
Description: Percentage of participants who progressed to death (all-cause mortality) was assessed.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

11. Secondary Outcome: Percentage of Participants Who Progressed to Respiratory Failure (of Any Cause) Requiring Mechanical Ventilation (Invasive or Noninvasive) Among Those Who Developed RSV LRTI or RSV-associated LRTC Per the EAC's Assessment
Description: Percentage of participants who progressed to respiratory failure (of any cause) requiring mechanical ventilation (invasive or noninvasive) among those who developed RSV LRTI or RSV-associated LRTC per the EAC's assessment was assessed. Here, '0' in the 'number of participants analyzed' field (N=0) signifies that no participants were available for the analysis because none of the participants developed RSV LRTI or RSV-associated LRTC per the EAC's Assessment.
Time Frame: Up to Day 49
Population: as for outcome 1
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of Participants Who Progressed to Respiratory Failure (of Any Cause) Requiring Mechanical Ventilation (Invasive or Noninvasive)
Description: Percentage of participants who progressed to respiratory failure (of any cause) requiring mechanical ventilation (invasive or noninvasive) was assessed.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

13. Secondary Outcome: Number of Supplemental Oxygen Free Days
Description: Number of supplemental oxygen free days was assessed. The number of supplemental oxygen free days was the number of days the participants did not receive/require supplemental oxygen during the first 28 days post treatment.
Time Frame: Through Day 28
Population: Efficacy analysis set included all participants who were randomized, treated (took at least 1 dose), and had a RSV infection confirmed by central laboratory analysis, excluding participants infected with a co-pathogen at baseline not identified during screening, analyzed as randomized. Here, "n" (number analyzed)" is defined as number of participants analyzed for each specified category.
Measure: Number; unit: Days
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Days
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 25
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 28
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 28

14. Secondary Outcome: Percentage of Participants With Treatment-emergent Oxygen Supplementation
Description: Percentage of participants who required treatment-emergent oxygen supplementation (e.g., supplemental oxygen, noninvasive pressure ventilation, invasive mechanical ventilation [tracheal tube, laryngeal mask or tracheostomy]). Any AE which occurred post first dose administration of study drug up to the end of study (that is, Day 49) were considered as treatment-emergent.
Time Frame: Up to Day 49
Population: Efficacy analysis set included all participants who were randomized, treated (took at least 1 dose), and had a RSV infection confirmed by central laboratory analysis, excluding participants infected with a co-pathogen at baseline not identified during screening, and were analyzed as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

15. Secondary Outcome: Respiratory Rate Over Time
Description: Respiratory rate over time was reported by investigator. In this outcome measure, only those timepoints in which individual participant had data were reported.
Time Frame: Baseline (Day 1), Days 15, 28, and 35
Population: The safety analysis set included all randomized participants who took at least 1 dose of study intervention and were analyzed 'as treated'. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represent number of participants with available data for each specified timepoint.
Measure: Number; unit: Breaths per minute
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 2
Breaths per minute
  Participant 1: Day 15: number analyzed (Participants) | 1
  Participant 1: Day 15 | 20
  Participant 1: Day 28: number analyzed (Participants) | 1
  Participant 1: Day 28 | 20
  Participant 1: Day 35: number analyzed (Participants) | 1
  Participant 1: Day 35 | 20
  Participant 2: Baseline: number analyzed (Participants) | 1
  Participant 2: Baseline | 16
  Participant 2: Day 15: number analyzed (Participants) | 1
  Participant 2: Day 15 | 20
  Participant 2: Day 28: number analyzed (Participants) | 1
  Participant 2: Day 28 | 16

16. Secondary Outcome: Heart Rate Over Time
Description: Heart rate over time was reported by investigator. In this outcome measure, only those timepoints in which individual participant had data were reported.
Time Frame: Baseline (Day 1), Days 15, 28, and 35
Population: The safety analysis set included all randomized participants who took at least 1 dose of study intervention and were analyzed 'as treated'. Here, 'n' (number analyzed) represent number of participants with available data for each specified timepoint.
Measure: Number; unit: Beats per minute
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Beats per minute
  Participant 1: Baseline: number analyzed (Participants) | 1
  Participant 1: Baseline | 83
  Participant 2: Baseline: number analyzed (Participants) | 1
  Participant 2: Baseline | 72
  Participant 2: Day 15: number analyzed (Participants) | 1
  Participant 2: Day 15 | 79
  Participant 2: Day 35: number analyzed (Participants) | 1
  Participant 2: Day 35 | 70
  Participant 3: Baseline: number analyzed (Participants) | 1
  Participant 3: Baseline | 70
  Participant 3: Day 15: number analyzed (Participants) | 1
  Participant 3: Day 15 | 73
  Participant 3: Day 28: number analyzed (Participants) | 1
  Participant 3: Day 28 | 78

17. Secondary Outcome: Peripheral Capillary Oxygen Saturation (SpO2) Over Time
Description: Peripheral capillary oxygen saturation (SpO2) over time was reported by investigator. In this outcome measure, only those timepoints in which individual participant had data were reported.
Time Frame: Baseline (Day 1), Days 15, 28, and 35
Population: as for outcome 16
Measure: Number; unit: Percentage (%) of Spo2
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage (%) of Spo2
  Participant 1: Baseline: number analyzed (Participants) | 1
  Participant 1: Baseline | 96
  Participant 2: Baseline: number analyzed (Participants) | 1
  Participant 2: Baseline | 98
  Participant 2: Day 15: number analyzed (Participants) | 1
  Participant 2: Day 15 | 97
  Participant 2: Day 28: number analyzed (Participants) | 1
  Participant 2: Day 28 | 100
  Participant 2: Day 35: number analyzed (Participants) | 1
  Participant 2: Day 35 | 96
  Participant 3: Baseline: number analyzed (Participants) | 1
  Participant 3: Baseline | 96
  Participant 3: Day 15: number analyzed (Participants) | 1
  Participant 3: Day 15 | 97
  Participant 3: Day 28: number analyzed (Participants) | 1
  Participant 3: Day 28 | 95

18. Secondary Outcome: Body Temperature Over Time
Description: Body temperature (in Degrees Celsius) over time was reported. In this outcome measure, only those timepoints in which individual participant had data were reported.
Time Frame: Baseline (Day 1), Days 15, 28, and 35
Population: as for outcome 16
Measure: Number; unit: Degree Celsius
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Degree Celsius
  Participant 1: Baseline: number analyzed (Participants) | 1
  Participant 1: Baseline | 36.3
  Participant 2: Baseline: number analyzed (Participants) | 1
  Participant 2: Baseline | 36.8
  Participant 2: Day 15: number analyzed (Participants) | 1
  Participant 2: Day 15 | 36.8
  Participant 2: Day 28: number analyzed (Participants) | 1
  Participant 2: Day 28 | 36.5
  Participant 2: Day 35 | 36.7
  Participant 3: Baseline: number analyzed (Participants) | 1
  Participant 3: Baseline | 35.9
  Participant 3: Day 15: number analyzed (Participants) | 1
  Participant 3: Day 15 | 36.1
  Participant 3: Day 28: number analyzed (Participants) | 1
  Participant 3: Day 28 | 36.2

19. Secondary Outcome: Percentage of Participants Hospitalized (of Participants Who Were Not Hospitalized at Baseline)
Description: Percentage of participants who were not hospitalized at baseline and required hospitalization during the study was assessed.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 0

20. Secondary Outcome: Percentage of Participants Who Were Re-hospitalized
Description: Percentage of participants who were re-hospitalized (of participants who were hospitalized at baseline and discharged during the study and of participants who were not hospitalized at baseline and required hospitalization and were discharged during the study) was assessed in this outcome measure.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Percentage of participants | 33.33

21. Secondary Outcome: Duration of Hospital Stay
Description: Duration (in days) of hospital stay was assessed.
Time Frame: Up to Day 49
Population: Efficacy analysis set included all participants who were randomized, treated (took at least 1 dose), and had a RSV infection confirmed by central laboratory analysis, excluding participants infected with a co-pathogen at baseline not identified during screening, analyzed as randomized. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Days
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 1
Days | 4

22. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: Duration of ICU stay was assessed. Duration (in hours) was defined as total number of hours a participant was in ICU from first dose of study drug until study termination.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Hours | 0 [0 to 0]

23. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 Treatment-emergent Adverse Events (TEAEs) in the Infections and Infestations System Organ Class
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE did not necessarily had a causal relationship with the intervention. Participants with Grade 3 or Grade 4 TEAE were assessed in this outcome measure. Any AE which occurred post first dose administration of study drug up to the end of study (that is, Day 49) were considered as treatment-emergent.
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Participants | 1

24. Secondary Outcome: Number of Participants With Respiratory Related AEs
Description: Number of participants with respiratory related AEs (respiratory infections) was assessed.
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Participants | 0

25. Secondary Outcome: Number of Participants With Thoracic-related AEs
Description: Number of participants with thoracic-related AEs was assessed.
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Participants | 0

26. Secondary Outcome: Number of Participants With Antibiotic Use Among Those Who Developed RSV LRTI or RSV-Associated LRTC Per the EAC's Assessment
Description: Number of participants with antibiotic use among those who developed RSV LRTI or RSV-associated LRTC per the EAC's assessment was assessed. Here, '0' in the 'number of participants analyzed' field (N=0) signifies that no participants were available for the analysis because none of the participants developed RSV LRTI or RSV-associated LRTC per the EAC's Assessment.
Time Frame: Up to Day 49
Population: as for outcome 1
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 0

27. Secondary Outcome: Plasma Concentration of JNJ-53718678
Description: Plasma Concentration of JNJ-53718678 was reported. In this outcome measure, only those timepoints in which individual participant had data were reported.
Time Frame: Days 1, 3, 8, 15 and 22
Population: PK analysis set included all participants who received JNJ-53718678 and for whom at least one PK concentration was reported. Here, 'n' (number analyzed) represents number of participants with available data for each specified timepoint.
Measure: Number; unit: Nanograms per milliliter (ng/mL)
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
Nanograms per milliliter (ng/mL)
  Participant 1: Day 1: number analyzed (Participants) | 1
  Participant 1: Day 1 | 1380
  Participant 2: Day 1: number analyzed (Participants) | 1
  Participant 2: Day 1 | 653
  Participant 2: Day 8: number analyzed (Participants) | 1
  Participant 2: Day 8 | 1780
  Participant 2: Day 15: number analyzed (Participants) | 1
  Participant 2: Day 15 | 1680
  Participant 2: Day 22: number analyzed (Participants) | 1
  Participant 2: Day 22 | 802
  Participant 3: Day 1: number analyzed (Participants) | 1
  Participant 3: Day 1 | 155
  Participant 3: Day 3: number analyzed (Participants) | 1
  Participant 3: Day 3 | 1680
  Participant 3: Day 8: number analyzed (Participants) | 1
  Participant 3: Day 8 | 2290
  Participant 3: Day 15: number analyzed (Participants) | 1
  Participant 3: Day 15 | 2510
  Participant 3: Day 22: number analyzed (Participants) | 1
  Participant 3: Day 22 | 812

28. Secondary Outcome: RSV Viral Load Over Time
Description: RSV viral load (RSV B) was measured over time by quantitative reverse transcription polymerase chain reaction (qRT-PCR) in the nasal swab specimens collected at the clinic visits and at home. In this outcome measure, only those timepoints in which individual participant had data were reported.
Time Frame: Baseline (Day 1), Days 15, 28, and 35
Population: Efficacy analysis set included all participants who were randomized, treated (took at least 1 dose), and had a RSV infection confirmed by central laboratory analysis, excluding participants infected with a co-pathogen at baseline not identified during screening, analyzed as randomized. Here, 'n' (number analyzed) represents number of participants with available data for each specified timepoint.
Measure: Number; unit: log10 copies per milliliter (mL)
Arm/Group | JNJ-53718678
Number analyzed (Participants) | 3
log10 copies per milliliter (mL)
  Participant 1: RSV B: Baseline: number analyzed (Participants) | 1
  Participant 1: RSV B: Baseline | 3.85
  Participant 1: RSV B: Day 28: number analyzed (Participants) | 1
  Participant 1: RSV B: Day 28 | 0
  Participant 2: RSV B: Baseline: number analyzed (Participants) | 1
  Participant 2: RSV B: Baseline | 8.01
  Participant 2: RSV B: Day 15: number analyzed (Participants) | 1
  Participant 2: RSV B: Day 15 | 5.95
  Participant 2: RSV B: Day 28: number analyzed (Participants) | 1
  Participant 2: RSV B: Day 28 | 5.16
  Participant 2: RSV B: Day 35: number analyzed (Participants) | 1
  Participant 2: RSV B: Day 35 | 5.63
  Participant 3: RSV B: Baseline: number analyzed (Participants) | 1
  Participant 3: RSV B: Baseline | 8.73
  Participant 3: RSV B: Day 15: number analyzed (Participants) | 1
  Participant 3: RSV B: Day 15 | 5.36
  Participant 3: RSV B: Day 28: number analyzed (Participants) | 1
  Participant 3: RSV B: Day 28 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 49
Description: The safety analysis set included all randomized participants who took at least 1 dose of study intervention and were analyzed 'as treated'.
Arm/Group | JNJ-53718678
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-53718678 (N=3)
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-53718678 (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cytomegalovirus Infection Reactivation (Infections and infestations) | 1
Dysgeusia (Nervous system disorders) | 1
Hot Flush (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
As the study was terminated early due to low number of participants enrolled, some efficacy analyses were not performed as per change in the planned analysis. Hence, data were collected and analyzed for safety and selected efficacy parameters only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT04056611/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT04056611/SAP_001.pdf